CLINICAL TRIAL: NCT01190969
Title: A Randomized Controlled Trial of Oral Nutritional Supplements on Nutritional Status and Clinical Outcomes in Malnourished Elderly
Brief Title: A Trial of Oral Nutritional Supplements on Nutritional Status and Clinical Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in recruiting elderly subjects
Sponsor: Singapore General Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GNSS 2010
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Malnutrition
Keywords: Elderly; malnutrition; nutritional supplement
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement (Ensure Plus) — Subjects will be provided with 2 to 3 serves of Ensure Plus (complete nutritional beverages) and to be taken between meals
  Other Names: Nutritional beverages

SUMMARY:
The purpose of this study is to determine whether short-term use of oral nutritional supplements as part of the diet improves nutritional and functional status of post-hospitalization malnourished elderly.

DETAILED DESCRIPTION:
Nutritional supplements have been shown to improve energy, protein, micronutrients intake, maintain or improve nutritional status in hospitalized malnourished elderly patients. However, its use in the elderly post-hospitalization is unknown, particularly in the local setting. This randomized controlled trial aims to investigate if provision of short term nutritional supplements to elderly malnourished patients after discharge from hospital improves nutritional status parameters. In addition, the impact of nutritional supplements on functional status, clinical outcome in terms of hospital readmission, number of visits to general practitioner/polyclinic and the acceptability of nutritional supplement in elderly are also examined. In this study, malnourished elderly subjects >65 years old identified by Malnutrition Universal Screening Tool from geriatric ward 63C will be recruited within 24 to 48 hours before discharge. They will be randomized into either intervention or control group. Subjects in the intervention group will receive nutritional supplements of 600 to 900 kcal as part of regular diet. As for the control group, these similar calories will be recommended from food fortification, as part of the standard care during diet counseling, to come from food. Both group subjects receive individualised assessment by the Dietitian. At baseline, nutritional status parameters such as weight, height, body mass index, skinfold thickness, handgrip strength, albumin and functional status will be measured. Subjects are then followed up at outpatient dietitian clinic 4 and 12 weeks from hospital discharge. Albumin test will be repeated at week 4 and week 12. They will keep a three-day food record end of week 1, week 4 and week 12 in order to assess their food and nutritional supplements intake. Compliance will be monitored from food diaries and interview. At the end of week 12, the same nutritional parameters will be re-evaluated for both groups. In addition, the number of hospital admissions, visits to the general practitioner/polyclinic and the acceptability of nutritional supplements will be determined. The results from this study will guide future nutritional interventions for the malnourished elderly post-hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 65 years old and to be discharged from Geriatric ward
* malnourished screened by Malnutrition Universal Screening Tool

Exclusion Criteria:

* are uncommunicative
* have a history of diabetes, chronic renal failure, liver disease
* are from long term residential homes like nursing homes
* incapable of taking study supplements to provide a minimum of 600 kcal/day as part of food intake
* intolerant to any of the ingredients in the study nutritional supplements
* require parenteral nutrition or enteral feeds as sole source of nutrition, e.g. patients who discharge home with tube feeding

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Body weight | Baseline, week 4 and week 12
  Body weight is measured to the nearest 0·01 kg using Seca clinical scales. If weight could not be measured accurately, recalled weight is used (Elia, 2003; Stratton et al. 2003a).

SECONDARY OUTCOMES:
Skinfold thickness | Baseline, week 4 and week 12
  Triceps skindfold thickness, mid arm circumference will be measured at above time points
Handgrip strength | Baseline, week 4 and week12
  Muscle grip strength will be measured at above time points
Blood Albumin | Baseline, week 4 and week12
Barthel Score | Baseline & week12
  Instrumental for assessing activities daily living
Number of visits to general practitioner/polyclinic | Week 12
  Above data will be collected at the end of the study
Hospital readmission | Week 12
  Above data will be collected at the end of the study
Acceptability of nutritional supplements | Week 12
  Above data will be collected at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Lee Boo Tan, BSc, MSc, Principal Investigator — Dietetics & Nutrition Services, Singapore General Hospital